CLINICAL TRIAL: NCT06998147
Title: Investigating Predictive Associations Among Postural Balance, Functional Mobility, Cognitive Function and Psychological Well-being in Patients With Multiple Sclerosis: A Cross-Sectional Study
Brief Title: Postural Control and Psychosocial Measures Associations in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azza Mohammed, Prof.Dr, Cairo University
Other Study IDs: No: H-02-J-002
Record Dates: First submitted 2025-05-19; First posted 2025-05-31 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Balance; Cognitive function; Depression; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Depression | interventions — Regression Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: correlation and regression analyses — to evaluate the association interplay among balance, functional mobility, cognitive function, psychological well-being, and community participation in addition to identify the anticipated contributing factors that function as predictors of MS features.

SUMMARY:
Balance deficits, gait abnormalities, impaired cognitive function, psychological disturbances and disconnection from community are key characteristics of multiple sclerosis (MS). Thus, exploring the interrelationships and the primary risk factors related to clinical manifestations and consequences of MS is of definite clinical significance. The primary aims of the study are to evaluate the association interplay among balance, functional mobility, cognitive function, psychological well-being, and community participation in addition to identify the anticipated contributing factors that function as predictors of MS features.

DETAILED DESCRIPTION:
This cross-sectional study will be carried out on sixty-four patients with MS. Balance performance was evaluated by a standardized Berg Balance Scale (BBS). Functional mobility will be measured via the well validated Timed Up and Go (TUG) test. Patients᾽ cognitive functions will be assessed by the Montreal Cognitive Assessment (MoCA), which is a sensitive screening test for the diagnosis of mild cognitive impairment. The psychological well-being will be measured based on the Hospital Anxiety and Depression Scale (HADS), which is widely employed to evaluate mood disturbances in clinical settings. Furthermore, community participation and engagement constraints will be measured with the Community Integration Questionnaire (CIQ) as they clearly capture the extent of functional and social integration into the community.

ELIGIBILITY:
Inclusion Criteria:

Participants will be screened for inclusion criteria to guarantee sample homogeneity and clinical applicability. First, all subjects will be diagnosed with MS confirmed by a neurologist according to the revised McDonald criteria. These criteria have the highest sensitivity and specificity and therefore are considered the gold standard in MS diagnosis. Second, participants will be be aged at least 18 years, so as to be able, cognitively and legally, to engage in the study as an informed study volunteer. Third, relapse- and relapse related treatments should be stopped by at least 1 month before the assessment. This is crucial in order to maximize the control of the transient influence of aggravation of the symptoms on patients᾽ cognitive and motor performance. Fourth, individuals will be eligible to participate in the study if they can ambulate, either independently or with the use of assistive device, as the study includes physical performance measures such as balance and gait. Finally, the maximum EDSS-value will be below 6 (moderate disability) to ensure independence of gait without constant support, as this is necessary to ensure comparability of balance and cognitive function.

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Sixty-four patients with MS will be recruited from the King Fahad General Hospital, a governmental hospital in Jeddah, Saudi Arabia. Full demographic data will be gathered and all subjects were carefully examined clinically. The study was ethically approved by the Institutional Review Board (IRB) of the Ministry of Health (MoH), Saudi Arabia (Approval No: H-02-J-002). A written informed consent of agreement to participate in the study will be obtained from all participants before enrollment and after being informed in detail about the purposes, study procedures, and their rights as research participants, in agreement with the ethical principles of the Declaration of Helsinki.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) scores | this outcome will take from 7 o 10 days to be completely assessed in all patients
  Balance performance was evaluated by a standardized Berg Balance Scale (BBS). scores ranges from 0 (no balance) to 54 (maximum balance)

SECONDARY OUTCOMES:
TUG test scores. | this outcome will take from 7 o 10 days to be completely assessed in all patients
  Functional mobility will be measured via the well validated Timed Up and Go (TUG) test.
Montreal Cognitive Assessment (MoCA) scores | this outcome will take from 5 to 7 days to be completely assessed in all patients
  Patients᾽ cognitive functions will be assessed by the Montreal Cognitive Assessment (MoCA)
HADS scores | this outcome will take from 5 to 7 days to be completely assessed in all patients
  The psychological well-being will be measured based on the Hospital Anxiety and Depression Scale (HADS). It consists of 14 items, divided into two subscales: 7 items for anxiety
CIQ scores | this outcome will take from 5 to 7 days to be completely assessed in all patients
  community participation and engagement constraints will be measured maximum total score of 30 points. A score of 26 or above is generally considered indicative of normal cognitive function. Scores between 18 and 25 suggest mild cognitive impairment, while scores from 10 to 17 indicate moderate cognitive impairment. A score below 10 reflects severe cognitive decline. According to MoCA guidelines, one point should be added to the total score for individuals with 12 years of education or less to account for the potential impact of educational background. Community Integration Questionnaire (CIQ)

CONTACTS AND LOCATIONS:
Overall Officials: Rasha M Hegazy, ph. D, Principal Investigator — Assistant professor of Neurology, Department of Physical Therapy for neurology and neurosurgery, Faculty of Physical Therapy, Cairo University, Giza, Egypt
Locations (1):
- Faculty of Physical Therapy, Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided